CLINICAL TRIAL: NCT00421941
Title: Use of a High-protein Enteral Formula Containing Prebiotics and Fish Oil in Critical Care
Brief Title: Enteral Feeding Study of Formula Containing Fish Oil in Critical Care Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet enrollment goal
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06.06.US.HCN
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Trauma; Tube Feeding
Keywords: enteral feeding; critical care; fish oil; surgical
MeSH Terms: conditions — Wounds and Injuries | interventions — Enteral Nutrition

INTERVENTIONS:
Procedure: Tube feeding

SUMMARY:
The purpose of this study is to evaluate the clinical applicability of an enteral tube feeding formula containing fish oil and prebiotics in a critical care population.

DETAILED DESCRIPTION:
In terms of nutrition support in the acute care setting, it is generally accepted that

1. earlier is better
2. enteral is superior to parenteral
3. the quality of nutrients appears more important than quantity
4. select populations will show additional benefit from specific nutrient supplementation.

The current study is designed to evaluate the tolerance of an enteral formula in trauma and surgery patients, as demonstrated by achieving and maintaining enteral feeding goal, gastrointestinal tolerance and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 70 years old
* New ICU admit
* Enteral tube feeding anticipated for at least 7 days
* Informed consent

Exclusion Criteria:

* Enteral tube feeding immediately prior to admit
* Parenteral feeding
* Medical condition that preclude receiving tube feeding or formula
* Determined by PI to be inappropriate
* Participating in another clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Clinical applicability as measured by the length of time between start of feeding to the first achievement of 800ml/day

SECONDARY OUTCOMES:
Gastrointestinal tolerance
Time to advance to full feed
Inflammatory markers
Infection

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martindale, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States